CLINICAL TRIAL: NCT06975098
Title: A Journey to Balance: Development and Validation of Individualized Life Balance Intervention for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Yun-Ling Chen, Assistant Professor, Chung Shan Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS2-23222
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Depression Disorders
Keywords: depression; life balance; individualized intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Life balance intervention group (Experimental): Intervention:
  A four-week individualized life balance intervention. The intervention combines weekly two-hour group sessions with telephone support provided 1-3 days prior to each session.
  Group session content is tailored to individual participant needs, identified through the Canadian Occupational Performance Measure (COPM) assessment.
  Interventions: Other: Life balance intervention group program

INTERVENTIONS:
Other: Life balance intervention group program — Life balance intervention group program is a four-week group intervention program for individuals with depression, with sessions lasting two hours each week. The program will address life balance issues such as daily scheduling, time management, stress coping, emotional regulation, and social participation, and will be tailored to individual patient needs. Through group discussions and practical exercises, participants will learn to apply these skills in their daily lives. Telephone support will be provided during the intervention period to offer emotional support and enhance participation rates.

SUMMARY:
The goal of this clinical intervention study is to enhance life balance in community-dwelling individuals with depression. The main question it aims to answer is:

Can an individualized life balance intervention, combining group sessions and telephone support, effectively improve life balance, time management, functional roles, quality of life, and reduce depression severity in individuals with depression?

Participants will:

Complete baseline assessments including demographics, illness-related information, and the Canadian Occupational Performance Measure (COPM).

Participate in four weekly, two-hour group sessions tailored to their individual needs identified through the COPM assessment.

Receive telephone support 1-3 days before each group session. Complete post-intervention assessments immediately after the four-week program and again one month later.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with depression by a psychiatrist.
* Assessed by a psychiatrist to be in a non-acute phase, approximately 4-8 weeks or more post-onset.
* Adults aged 20 or above with independent behavioral capacity.
* Literate, with basic cognitive function.

Exclusion Criteria:

* Diagnosis of schizophrenia spectrum and other psychotic disorders, bipolar and related disorders, substance-related and addictive disorders, neurodevelopmental disorders, neurocognitive disorders, or substance/medication-induced depressive disorders.
* Significant physical illnesses requiring active and long-term treatment, such as cancer, cerebrovascular disease (stroke), spinal cord injury, congenital or genetic diseases, chronic renal failure, systemic autoimmune diseases, or burns.
* Lack of willingness to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (baseline) | baseline
  The Canadian Occupational Performance Measure (COPM) is a client-centered assessment tool used to evaluate changes in the performance and satisfaction of an individual's perceived occupational performance problems over time. When occupational performance is difficult to quantify, the COPM serves as an outcome measure. Therapists conduct a semi-structured interview with the individual to identify their most important occupational performance problems, and then rate the importance, performance, and satisfaction of each problem on a scale of 1 to 10. Higher scores indicate greater importance, performance, and satisfaction. During reassessment, individuals re-rate these occupational performance problems. A change of 2 points or more between initial and subsequent scores is considered clinically significant.
Canadian Occupational Performance Measure (post-intervention) | post-intervention (up to 4 weeks)
  The Canadian Occupational Performance Measure (COPM) is a client-centered assessment tool used to evaluate changes in the performance and satisfaction of an individual's perceived occupational performance problems over time. When occupational performance is difficult to quantify, the COPM serves as an outcome measure. Therapists conduct a semi-structured interview with the individual to identify their most important occupational performance problems, and then rate the importance, performance, and satisfaction of each problem on a scale of 1 to 10. Higher scores indicate greater importance, performance, and satisfaction. During reassessment, individuals re-rate these occupational performance problems. A change of 2 points or more between initial and subsequent scores is considered clinically significant.
Canadian Occupational Performance Measure (follow-up) | 1-month follow-up
  The Canadian Occupational Performance Measure (COPM) is a client-centered assessment tool used to evaluate changes in the performance and satisfaction of an individual's perceived occupational performance problems over time. When occupational performance is difficult to quantify, the COPM serves as an outcome measure. Therapists conduct a semi-structured interview with the individual to identify their most important occupational performance problems, and then rate the importance, performance, and satisfaction of each problem on a scale of 1 to 10. Higher scores indicate greater importance, performance, and satisfaction. During reassessment, individuals re-rate these occupational performance problems. A change of 2 points or more between initial and subsequent scores is considered clinically significant.
Occupational balance (baseline) | baseline
  Occupational Balance Questionnaire 11-Chinese version (OBQ11-C) is a 11-item questionnaire with a four point rating scale for each item (from 0 to 3) by the level of agreemtent with each of the affirmations. The OBQ11-C is used to measure the perception of current occupational balance in daily life. The total score is ranged from 0 to 33. A higher score indicates a greater occupational balance.
Occupational balance (post-intervention) | post-intervention (up to 4 weeks)
  Occupational Balance Questionnaire 11-Chinese version (OBQ11-C) is a 11-item questionnaire with a four point rating scale for each item (from 0 to 3) by the level of agreemtent with each of the affirmations. The OBQ11-C is used to measure the perception of current occupational balance in daily life. The total score is ranged from 0 to 33. A higher score indicates a greater occupational balance.
Occupational balance (follow-up) | 1-month follow-up
  Occupational Balance Questionnaire 11-Chinese version (OBQ11-C) is a 11-item questionnaire with a four point rating scale for each item (from 0 to 3) by the level of agreemtent with each of the affirmations. The OBQ11-C is used to measure the perception of current occupational balance in daily life. The total score is ranged from 0 to 33. A higher score indicates a greater occupational balance.
Occupational questionnaire (baseline) | baseline
  Occupational questionnaire (OQ) is used to record daily occupations on 30-minute interval for a typical day. Each activity need to be classified as work, activity of daily living, recreation or rest and be rated for the competence, value, and interest using a five point rating scale. It indicates how well the participants do the activity, how important the activity is as well as how enjoyable the activity is. The higher score means better satisfaction, value and enjoyment of activity that the participant did.
Occupational questionnaire (post-intervention) | post-intervention (up to 4 weeks)
  Occupational questionnaire (OQ) is used to record daily occupations on 30-minute interval for a typical day. Each activity need to be classified as work, activity of daily living, recreation or rest and be rated for the competence, value, and interest using a five point rating scale. It indicates how well the participants do the activity, how important the activity is as well as how enjoyable the activity is. The higher score means better satisfaction, value and enjoyment of activity that the participant did.
Occupational questionnaire (follow-up) | 1-month follow-up
  Occupational questionnaire (OQ) is used to record daily occupations on 30-minute interval for a typical day. Each activity need to be classified as work, activity of daily living, recreation or rest and be rated for the competence, value, and interest using a five point rating scale. It indicates how well the participants do the activity, how important the activity is as well as how enjoyable the activity is. The higher score means better satisfaction, value and enjoyment of activity that the participant did.
Role checklist (baseline) | baseline
  Role checklist is used to assess the major roles that organize participant's daily life and the value of each role. The roles included the student, worker, volunteer, caregiver, home maintainer, friend, family member, religious participant, hobbyist, and participant in organizations. A higher number of roles means participating more roles in daily life. A higher score in the value of roles means more productive behaviors participants needed or desired.
Role checklist (post-intervention) | post-intervention (up to 4 weeks)
  Role checklist is used to assess the major roles that organize participant's daily life and the value of each role. The roles included the student, worker, volunteer, caregiver, home maintainer, friend, family member, religious participant, hobbyist, and participant in organizations. A higher number of roles means participating more roles in daily life. A higher score in the value of roles means more productive behaviors participants needed or desired.
Role checklist (follow-up) | 1-month follow-up
  Role checklist is used to assess the major roles that organize participant's daily life and the value of each role. The roles included the student, worker, volunteer, caregiver, home maintainer, friend, family member, religious participant, hobbyist, and participant in organizations. A higher number of roles means participating more roles in daily life. A higher score in the value of roles means more productive behaviors participants needed or desired.

SECONDARY OUTCOMES:
Quality of life (baseline) | baseline
  The World Health Organization Quality of Life Questionnaire- BREF Taiwan version (WHOQOL-BREF-TW) is a 28-item self-report questionnaire with a five point rating scale for each item (from 1 to 5). There are four domains in WHOQOL-BREF-TW, including physical health, psychological health, social relationships, and environment. A higher score indicates a higher quality of life.
Quality of life (post-intervention) | post-intervention (up to 4 weeks)
  The World Health Organization Quality of Life Questionnaire- BREF Taiwan version (WHOQOL-BREF-TW) is a 28-item self-report questionnaire with a five point rating scale for each item (from 1 to 5). There are four domains in WHOQOL-BREF-TW, including physical health, psychological health, social relationships, and environment. A higher score indicates a higher quality of life.
Quality of life (follow-up) | 1-month follow-up
  The World Health Organization Quality of Life Questionnaire- BREF Taiwan version (WHOQOL-BREF-TW) is a 28-item self-report questionnaire with a five point rating scale for each item (from 1 to 5). There are four domains in WHOQOL-BREF-TW, including physical health, psychological health, social relationships, and environment. A higher score indicates a higher quality of life.
Depression (baseline) | baseline
  Beck Depression Inventory - II (BDI-II) contains 21 items (each of them is scored on a scale of 0-3) in order to measure the depressive symptoms of participants. Higher scores indicates greater level of depression. 0-13 is considered a none or minimal, 14-19 is mild, 20-28 is moderate, and 29-63 is severe level of depression.
Depression (post-intervention) | post-intervention (up to 4 weeks)
  Beck Depression Inventory - II (BDI-II) contains 21 items (each of them is scored on a scale of 0-3) in order to measure the depressive symptoms of participants. Higher scores indicates greater level of depression. 0-13 is considered a none or minimal, 14-19 is mild, 20-28 is moderate, and 29-63 is severe level of depression.
Depression (follow-up) | 1-month follow-up
  Beck Depression Inventory - II (BDI-II) contains 21 items (each of them is scored on a scale of 0-3) in order to measure the depressive symptoms of participants. Higher scores indicates greater level of depression. 0-13 is considered a none or minimal, 14-19 is mild, 20-28 is moderate, and 29-63 is severe level of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yao G, Chung CW, Yu CF, Wang JD. Development and verification of validity and reliability of the WHOQOL-BREF Taiwan version. J Formos Med Assoc. 2002 May;101(5):342-51. PMID 12101852
- [Result] World Health Organization. (2017). Depression and Other Common Mental Disorders: Global Health Estimates. World Health Organization (Licence: CC BY-NC-SA 3.0 IGO). http://www.who.int/mental_health/management/depression/prevalence_global_health_estimates/en/
- [Result] Wagman P, Hakansson C, Bjorklund A. Occupational balance as used in occupational therapy: a concept analysis. Scand J Occup Ther. 2012 Jul;19(4):322-7. doi: 10.3109/11038128.2011.596219. Epub 2011 Jul 25. PMID 21780985
- [Result] Wagman P, Hjarthag F, Hakansson C, Hedin K, Gunnarsson AB. Factors associated with higher occupational balance in people with anxiety and/or depression who require occupational therapy treatment. Scand J Occup Ther. 2021 Aug;28(6):426-432. doi: 10.1080/11038128.2019.1693626. Epub 2019 Dec 14. PMID 31838931
- [Result] Wagman P, Hakansson C. Introducing the Occupational Balance Questionnaire (OBQ). Scand J Occup Ther. 2014 May;21(3):227-31. doi: 10.3109/11038128.2014.900571. Epub 2014 Mar 21. PMID 24649971
- [Result] Uyeshiro Simon A, Collins CER. Lifestyle Redesign(R) for Chronic Pain Management: A Retrospective Clinical Efficacy Study. Am J Occup Ther. 2017 Jul/Aug;71(4):7104190040p1-7104190040p7. doi: 10.5014/ajot.2017.025502. PMID 28661383
- [Result] Smith NR, Kielhofner G, Watts JH. The relationships between volition, activity pattern, and life satisfaction in the elderly. Am J Occup Ther. 1986 Apr;40(4):278-83. doi: 10.5014/ajot.40.4.278. PMID 3963137
- [Result] Skjutar A, Schult ML, Christensson K, Mullersdorf M. Indicators of need for occupational therapy in patients with chronic pain: occupational therapists' focus groups. Occup Ther Int. 2010 Jun;17(2):93-103. doi: 10.1002/oti.282. PMID 19653210
- [Result] Shang, C. Y., Liao, S. C., & Lee, M. B. (2003). Trends of visiting rate of depressive outpatients in psychiatric clinic. Formosan Journal of Medicine, 7(4), 502-509. (in Chinese).
- [Result] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Result] Pyatak E, King M, Vigen CLP, Salazar E, Diaz J, Schepens Niemiec SL, Blanchard J, Jordan K, Banerjee J, Shukla J. Addressing Diabetes in Primary Care: Hybrid Effectiveness-Implementation Study of Lifestyle Redesign(R) Occupational Therapy. Am J Occup Ther. 2019 Sep/Oct;73(5):7305185020p1-7305185020p12. doi: 10.5014/ajot.2019.037317. PMID 31484021
- [Result] Peral-Gomez P, Lopez-Roig S, Pastor-Mira MA, Abad-Navarro E, Valera-Gran D, Hakansson C, Wagman P. Cultural Adaptation and Psychometric Properties of the Spanish Version of the Occupational Balance Questionnaire: An Instrument for Occupation-Based Research. Int J Environ Res Public Health. 2021 Jul 14;18(14):7506. doi: 10.3390/ijerph18147506. PMID 34299957
- [Result] Mcmullen C, Liu L, Bulkley JE, Hornbrook MC, Wendel C, Grant M, Altschuler A, Temple LK, Krouse RS, Herrinton L. Participation in Activities Associated With Quality of Life for Long-Term Survivors of Rectal Cancer. Perm J. 2017;21:16-011. doi: 10.7812/TPP/16-011. PMID 28241904
- [Result] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Result] Magnusson L, Hakansson C, Brandt S, Oberg M, Orban K. Occupational balance and sleep among women. Scand J Occup Ther. 2021 Nov;28(8):643-651. doi: 10.1080/11038128.2020.1721558. Epub 2020 Mar 18. PMID 32186421
- [Result] Maeir T, Beit-Yosef A, Wechsler T, Safra Y, Zilbershlag Y, Katz N, Gilboa Y. The Feasibility and Efficacy of an Israeli Lifestyle Redesign(R)-Based Program for Well Older Adults: A Pilot Study. OTJR (Thorofare N J). 2021 Jan;41(1):47-55. doi: 10.1177/1539449220928141. Epub 2020 Jun 21. PMID 32567478
- [Result] Lund K, Hultqvist J, Bejerholm U, Argentzell E, Eklund M. Group leader and participant perceptions of Balancing Everyday Life, a group-based lifestyle intervention for mental health service users. Scand J Occup Ther. 2020 Aug;27(6):462-473. doi: 10.1080/11038128.2018.1551419. Epub 2019 Feb 1. PMID 30706746
- [Result] Lund K, Argentzell E, Bejerholm U, Eklund M. Breaking a cycle of perceived failure: The process of making changes toward a more balanced lifestyle. Aust Occup Ther J. 2019 Oct;66(5):627-636. doi: 10.1111/1440-1630.12604. Epub 2019 Jul 25. PMID 31344759
- [Result] Lund A, Michelet M, Sandvik L, Wyller T, Sveen U. A lifestyle intervention as supplement to a physical activity programme in rehabilitation after stroke: a randomized controlled trial. Clin Rehabil. 2012 Jun;26(6):502-12. doi: 10.1177/0269215511429473. Epub 2011 Dec 14. PMID 22169830
- [Result] Lin EC, Chan CH, Shao WC, Lin MF, Shiau S, Mueser KT, Huang SC, Wang HS. A randomized controlled trial of an adapted Illness Management and Recovery program for people with schizophrenia awaiting discharge from a psychiatric hospital. Psychiatr Rehabil J. 2013 Dec;36(4):243-9. doi: 10.1037/prj0000013. PMID 24320832
- [Result] Liao SC, Chen WJ, Lee MB, Lung FW, Lai TJ, Liu CY, Lin CY, Yang MJ, Chen CC. Low prevalence of major depressive disorder in Taiwanese adults: possible explanations and implications. Psychol Med. 2012 Jun;42(6):1227-37. doi: 10.1017/S0033291711002364. Epub 2011 Nov 4. PMID 22051196
- [Result] Lagueux E, Masse J, Levasseur M, Page R, Depelteau A, Levesque MH, Tousignant-Laflamme Y, Pinard AM. Pilot Study of French-Canadian Lifestyle Redesign(R) for Chronic Pain Management. OTJR (Thorofare N J). 2021 Apr;41(2):80-89. doi: 10.1177/1539449220982908. Epub 2021 Jan 3. PMID 33393417
- [Result] Krupa, T., Kirsh, B., Pitts, D., & Fossey, E. (2016). Bruce & Borg's Psychosocial Frames of Reference: Theories, Models and Approaches for Occupation-Based Practice (4th ed.). Slack.
- [Result] Johansson C, Isaksson G. Experiences of participation in occupations of women on long-term sick leave. Scand J Occup Ther. 2011 Dec;18(4):294-301. doi: 10.3109/11038128.2010.521950. Epub 2010 Oct 21. PMID 20961264
- [Result] Jakobsen K, Magnus E, Lundgren S, Reidunsdatter RJ. Everyday life in breast cancer survivors experiencing challenges: A qualitative study. Scand J Occup Ther. 2018 Jul;25(4):298-307. doi: 10.1080/11038128.2017.1335777. Epub 2017 May 31. PMID 28562163
- [Result] Hultqvist J, Lund K, Argentzell E, Eklund M. Predictors of clinically important improvements in occupational and quality of life outcomes among mental health service users after completion and follow-up of a lifestyle intervention: multiple regression modelling based on longitudinal data. BMC Psychol. 2019 Dec 17;7(1):83. doi: 10.1186/s40359-019-0359-z. PMID 31847910
- [Result] Huang CY, Sousa VD, Tsai CC, Hwang MY. Social support and adaptation of Taiwanese adults with mental illness. J Clin Nurs. 2008 Jul;17(13):1795-802. doi: 10.1111/j.1365-2702.2008.02310.x. PMID 18578782
- [Result] Hakansson C, Wagman P, Hagell P. Construct validity of a revised version of the Occupational Balance Questionnaire. Scand J Occup Ther. 2020 Aug;27(6):441-449. doi: 10.1080/11038128.2019.1660801. Epub 2019 Sep 14. PMID 31524026
- [Result] Gunnarsson, B. (2008). The Tree Theme Method-An Occupational Therapy Intervention Applied in Outpatient Psychiatric Care (Vol. 2008). Lund University.
- [Result] Gunnarsson AB, Wagman P, Hakansson C, Hedin K. The Tree Theme Method(R) (TTM), an occupational therapy intervention for treating depression and anxiety: study protocol of a randomized controlled trial. BMC Psychol. 2015 Nov 9;3:40. doi: 10.1186/s40359-015-0097-9. PMID 26552426
- [Result] Gunnarsson AB, Jansson JA, Eklund M. The Tree Theme Method in psychosocial occupational therapy: a case study. Scand J Occup Ther. 2006 Dec;13(4):229-40. doi: 10.1080/11038120600772908. PMID 17203673
- [Result] Gunnarsson AB, Hakansson C, Hedin K, Wagman P. Outcomes of the Tree Theme Method versus regular occupational therapy: A longitudinal follow-up. Aust Occup Ther J. 2022 Aug;69(4):379-390. doi: 10.1111/1440-1630.12796. Epub 2022 Mar 7. PMID 35257386
- [Result] Gunnarsson AB, Eklund M. The Tree Theme Method as an intervention in psychosocial occupational therapy: client acceptability and outcomes. Aust Occup Ther J. 2009 Jun;56(3):167-76. doi: 10.1111/j.1440-1630.2008.00738.x. PMID 20854510
- [Result] GBD 2019 Mental Disorders Collaborators. Global, regional, and national burden of 12 mental disorders in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Psychiatry. 2022 Feb;9(2):137-150. doi: 10.1016/S2215-0366(21)00395-3. Epub 2022 Jan 10. PMID 35026139
- [Result] Eklund M, Tjornstrand C, Sandlund M, Argentzell E. Effectiveness of Balancing Everyday Life (BEL) versus standard occupational therapy for activity engagement and functioning among people with mental illness - a cluster RCT study. BMC Psychiatry. 2017 Nov 9;17(1):363. doi: 10.1186/s12888-017-1524-7. PMID 29121882
- [Result] Eklund M, Orban K, Argentzell E, Bejerholm U, Tjornstrand C, Erlandsson LK, Hakansson C. The linkage between patterns of daily occupations and occupational balance: Applications within occupational science and occupational therapy practice. Scand J Occup Ther. 2017 Jan;24(1):41-56. doi: 10.1080/11038128.2016.1224271. Epub 2016 Aug 30. PMID 27575654
- [Result] Eklund M, Lund K, Argentzell E. The impact of the BEL intervention on levels of motivation, engagement and recovery in people who attend community mental health services. Scand J Occup Ther. 2023 Aug;30(6):862-872. doi: 10.1080/11038128.2023.2184717. Epub 2023 Mar 3. PMID 36867590
- [Result] Eklund M, Leufstadius C, Bejerholm U. Time use among people with psychiatric disabilities: implications for practice. Psychiatr Rehabil J. 2009 Winter;32(3):177-91. doi: 10.2975/32.3.2009.177.191. PMID 19136350
- [Result] Eklund M, Brunt D, Argentzell E. Perceived occupational balance and well-being among people with mental illness living in two types of supported housing. Scand J Occup Ther. 2020 Aug;27(6):450-461. doi: 10.1080/11038128.2019.1622771. Epub 2019 Jun 7. PMID 31170857
- [Result] Eklund M, Argentzell E. Perception of occupational balance by people with mental illness: A new methodology. Scand J Occup Ther. 2016 Jul;23(4):304-13. doi: 10.3109/11038128.2016.1143529. Epub 2016 Feb 12. PMID 26872496
- [Result] Crist, P. H., Davis, C. G., & Coffin, P. S. (2000). The effects of employment and mental health status on the balance of work, play/leisure, self-care, and rest. Occupational Therapy in Mental Health, 15(1), 27-42. https://doi.org/10.1300/J004v15n01_02
- [Result] Chen YL, Pan AW, Hsiung PC, Chung L, Lai JS, Shur-Fen Gau S, Chen TJ. Life Adaptation Skills Training (LAST) for persons with depression: A randomized controlled study. J Affect Disord. 2015 Oct 1;185:108-14. doi: 10.1016/j.jad.2015.06.022. Epub 2015 Jun 27. PMID 26162281
- [Result] Chen, H. (2000). Manual for the Beck Depression Inventory-II (Chinese version). Chinese Behavioural Science Corporation.
- [Result] Carswell A, McColl MA, Baptiste S, Law M, Polatajko H, Pollock N. The Canadian Occupational Performance Measure: a research and clinical literature review. Can J Occup Ther. 2004 Oct;71(4):210-22. doi: 10.1177/000841740407100406. PMID 15586853
- [Result] Brown, C., Stoffel, V. C., & Muňoz, J. P. (2019). Occupational Therapy in Mental Health: A Vision for Participation (2nd ed.). F.A. Davis. .
- [Result] Birgitta Gunnarsson A, Wagman P, Hedin K, Hakansson C. Treatment of depression and/or anxiety - outcomes of a randomised controlled trial of the tree theme method(R) versus regular occupational therapy. BMC Psychol. 2018 May 23;6(1):25. doi: 10.1186/s40359-018-0237-0. PMID 29792226
- [Result] Bakish D. New standard of depression treatment: remission and full recovery. J Clin Psychiatry. 2001;62 Suppl 26:5-9. PMID 11775091
- [Result] Occupational Therapy Practice Framework: Domain and Process-Fourth Edition. Am J Occup Ther. 2020 Aug 1;74(Supplement_2):7412410010p1-7412410010p87. doi: 10.5014/ajot.2020.74S2001. PMID 34780625